CLINICAL TRIAL: NCT03289533
Title: AN OPEN LABEL, SINGLE ARM PHASE 1B STUDY OF AVELUMAB PLUS AXITINIB AS FIRST LINE TREATMENT IN PATIENTS WITH ADVANCED HEPATOCELLULAR CARCINOMA
Brief Title: A Study Of Avelumab In Combination With Axitinib In Advanced HCC (VEGF Liver 100)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B9991024
Record Dates: First submitted 2017-08-28; First posted 2017-09-21 (Actual); Results first posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Cancer; Hepatocellular carcinoma; Liver disease; Avelumab; Axitinib
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasms; Liver Diseases | interventions — avelumab; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental 1 (Experimental): Avelumab (MSB0010718C) in combination with axitinib (AG-013736)
  Interventions: Drug: Avelumab (MSB0010718C); Drug: Axitinib (AG-013736)

INTERVENTIONS:
Drug: Avelumab (MSB0010718C) — Patients will receive avelumab 10 mg/kg Q2W in combination with axitinib 5 mg BID.
Drug: Axitinib (AG-013736) — Patients will receive avelumab 10 mg/kg Q2W in combination with axitinib 5 mg BID.

SUMMARY:
To evaluate the safety, efficacy and PK of avelumab in combination with axitinib as first line treatment in patients with advanced HCC

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of locally advanced or metastatic HCC, obtained by histology/cytology (on a prior tumor biopsy) or by imaging with serum α-fetoprotein (AFP) ≥400 ng/mL.
* All patients must provide at least 1 archival tumor specimen. If archival tumor specimen is no longer available, de novo tumor biopsy will be required during screening.
* HCC not amenable to local therapy.
* Measurable disease according to RECIST v. 1.1.
* Child Pugh Class A disease.
* BCLC stage B or C disease.
* No evidence of uncontrolled hypertension as documented by 2 baseline blood pressure readings taken at least 1 hour apart.
* ECOG performance status 0 or 1.
* Adequate bone marrow function, renal and liver functions
* Left ventricular ejection fraction (LVEF) ≥ lower limit of normal (LLN) as assessed by multigated acquisition (MUGA) scan or echocardiogram (ECHO).

Exclusion Criteria:

* Prior systemic treatment for advanced HCC, including prior treatment with approved or investigational drugs.
* Any prior locoregional therapy within 4 weeks and radiotherapy or surgical procedure within 2 weeks (4 weeks for major surgery) of enrollment.
* Patients with known symptomatic brain metastases requiring steroids.
* Presence of hepatic encephalopathy (ie, Child Pugh score of 2 or 3) and/or clinically relevant ascites (ie, Child Pugh score of 3).
* Presence of main portal vein invasion by HCC.
* Any of the following within the 12 months prior to enrollment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, LVEF less than LLN, clinically significant pericardial effusion, cerebrovascular accident, transient ischemic attack.
* Active infection requiring systemic therapy except for hepatitis C virus (HCV) and hepatitis B virus (HBV).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- Japan (7):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Iizuka Hospital, Iizuka, Fukuoka
  - Kindai University Hospital, Department of Gastroenterology and Hepatology, Ōsaka-sayama, Osaka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Kyorin University Hospital, Department of Medical Oncology, Mitaka-shi, Tokyo
  - Japanese Red Cross Musashino Hospital, Musashino, Tokyo
  - National Hospital Organization Kyushu Medical Center, Fukuoka

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B9991024

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with advanced hepatocellular carcinoma (HCC) who did not receive any prior systemic therapy were enrolled in this study.
Groups:
- Avelumab + Axitinib: Participants with advanced HCC were administered with Avelumab 10 milligram per kilogram (mg/kg) as 1-hour intravenous (IV) infusion, on Day 1 of each cycle along with Axitinib 5 milligram (mg) oral tablets, twice daily on a continuous dosing schedule (without a break in dosing except in case of drug-related toxicity) until disease progression, participant refusal, unacceptable toxicity, lost to follow-up, or until study termination by the sponsor, whichever occurred first (up to maximum of 40 cycles). Duration of each cycle =14 days.
Period: Overall Study
Arm/Group | Avelumab + Axitinib
Started | 22
Completed | 0
Not Completed | 22
Not completed — Death | 12
Not completed — Terminated from study by sponsor | 10

BASELINE CHARACTERISTICS:
Population: Full analysis set included participants who received at least one dose of study drug.
Groups:
- Avelumab + Axitinib: Participants with advanced HCC were administered with Avelumab 10 mg/kg as 1-hour IV infusion, on Day 1 of each cycle along with Axitinib 5 mg oral tablets, twice daily on a continuous dosing schedule (without a break in dosing except in case of drug-related toxicity) until disease progression, participant refusal, unacceptable toxicity, lost to follow-up, or until study termination by the sponsor, whichever occurred first (up to maximum of 40 cycles). Duration of each cycle =14 days.
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (14.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 22
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) by Severity as Graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version (v.) 4.03
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AEs were graded by investigator according to NCI CTCAE v.4.03 as follows: Grade 1: mild AE, Grade 2: moderate AE, Grade 3: severe AE, Grade 4: life-threatening consequences and urgent intervention indicated, Grade 5: death related to AE.
Time Frame: From first dose of study drug up to 30 days after last dose of study drug or initiation of new anti-cancer drug therapy, whichever occurred first (maximum up to 21 months)
Population: Safety analysis set included participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 22
Participants
  Grade 1 | 2
  Grade 2 | 3
  Grade 3 | 16
  Grade 4 | 1
  Grade 5 | 0

2. Primary Outcome: Number of Participants With Abnormal Laboratory Parameter Values (Hematology) as Graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Event (CTCAE) Version 4.03
Description: As per NCI-CTCAE v 4.03, anemia Grade 1= Less than (<) lower limit of normal (LLN) to 100 gram per liter (g/L),Grade 2= <100 to 80 g/L; hemoglobin increased: Grade 1= increase of greater than (>) 0 to 2 gram per deciliter(g/dL) above upper limit of normal [ULN]; lymphocyte count decreased: Grade 1= <LLN to 0.8*10^9/L, Grade 2= <0.8*10^9/L to 0.5*10^9/L, Grade 3= <0.5*10^9/L to 0.2*10^9/L ; lymphocyte count increased: Grade 2= >4*10^9/L to 20*10^9/L; neutrophil count decreased: Grade 1= <LLN to 1.5*10^9/L ,Grade 2= <1.5*10^9/L to 1.0*10^9/L; platelet count decreased: Grade 1= <LLN to 75.0*10^9/L, Grade 2= <75.0*10^9/L to 50.0*10^9/L; white blood cell decreased: Grade 1= <LLN to 3*10^9/L, Grade 2= <3*10^9/L to 2*10^9/L.
Time Frame: as for outcome 1
Population: Safety analysis set included participants who received at least one dose of study drug. Categories with at least 1 participant with abnormality were reported in this outcome measure. One participant might have more than 1 abnormality.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 22
Participants
  Anemia: Grade 1 | 13
  Anemia: Grade 2 | 3
  Hemoglobin increased: Grade 1 | 5
  Lymphocyte count decreased: Grade 1 | 11
  Lymphocyte count decreased: Grade 2 | 2
  Lymphocyte count decreased: Grade 3 | 1
  Lymphocyte count increased: Grade 2 | 1
  Neutrophil count decreased: Grade 1 | 3
  Neutrophil count decreased: Grade 2 | 5
  Platelet count decreased: Grade 1 | 14
  Platelet count decreased: Grade 2 | 2
  White blood cell decreased: Grade 1 | 1
  White blood cell decreased: Grade 2 | 4

3. Primary Outcome: Number of Participants With Abnormal Laboratory Parameter Values (Chemistry) as Graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Event (CTCAE) Version (v) 4.03
Description: ALT,ALP,AST increased grades(g):g1>ULN-3.0*ULN,g2>3.0-5.0*ULN,g3>5.0-20.0*ULN; blood bilirubin increased:g1>ULN-1.5*ULN, g2>1.5-3.0*ULN, g3>3.0-10.0*ULN; [cholesterol high:g1>ULN-7.75, g2 >7.75-10.34,g4 >12.92]millimoles per liter(mmol/L);creatine phosphokinase, gamma-glutamyl transferase(ggt) increased g1>ULN-2.5*ULN, g2>2.5*ULN-5*ULN; Ggt increased g3 >5.0-20.0*ULN; Creatinine increased: g1>ULN-1.5*ULN; [hypoalbuminemia:g1<LLN-30,g2<30-20] grams per liter(g/L);[hyperglycemia:g1> ULN-8.9,g2> 8.9-13.9,g3> 13.9-27.8;hypermagnesemia:g1>ULN-1.23;hypercalcemia:g1>ULN -2.9;hyperkalemia:g1>ULN-5.5,hypernatremia:g1>ULN-150;hypertriglyceridemia g1:1.71-3.42,g2 >3.42-5.7;hypocalcemia:g1<LLN-2.0,hypoglycemia:g1<LLN-3.0, g2<3.0-2.2;hypokalemia:g2<LLN-3.0,g4<2.5,hypomagnesemia:g1<LLN-0.5,hyponatremia:g1<LLN-130, g3<130-120,hypophosphatemia:g1<LLN-0.8,g2<0.8-0.6]mmol/L;lipase increased:g1>ULN-1.5*ULN,g3 >2.0-5.0*ULN;serum amylase increased:g1>ULN-1.5*ULN, g2>1.5-2.0*ULN,g3>2.0-5.0*ULN.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 22
Participants
  Alanine aminotransferase (ALT) increased: Grade 1 | 15
  ALT increased: Grade 2 | 2
  ALT increased: Grade 3 | 1
  Alkaline phosphatase (ALP) increased: Grade 1 | 11
  ALP increased: Grade 2 | 2
  ALP increased: Grade 3 | 3
  Aspartate aminotransferase(AST) increased: Grade 1 | 15
  AST increased: Grade 2 | 4
  AST increased: Grade 3 | 2
  Blood bilirubin increased: Grade 1 | 4
  Blood bilirubin increased: Grade 2 | 2
  Blood bilirubin increased: Grade 3 | 1
  Cholesterol high: Grade 1 | 5
  Cholesterol high: Grade 2 | 1
  Cholesterol high: Grade 4 | 1
  Creatine phosphokinase increased: Grade 1 | 2
  Creatine phosphokinase increased: Grade 2 | 1
  Creatinine increased: Grade 1 | 21
  Gamma-glutamyl transferase(Ggt) increased: Grade 1 | 6
  Ggt increased: Grade 2 | 5
  Ggt increased: Grade 3 | 7
  Hypercalcemia: Grade 1 | 10
  Hyperglycemia: Grade 1 | 11
  Hyperglycemia: Grade 2 | 2
  Hyperglycemia: Grade 3 | 1
  Hyperkalemia: Grade 1 | 4
  Hypermagnesemia: Grade 1 | 4
  Hypernatremia: Grade 1 | 3
  Hypertriglyceridemia; Grade 1 | 9
  Hypertriglyceridemia; Grade 2 | 3
  Hypoalbuminemia: Grade 1 | 15
  Hypoalbuminemia: Grade 2 | 3
  Hypocalcemia: Grade 1 | 1
  Hypoglycemia: Grade 1 | 2
  Hypoglycemia: Grade 2 | 1
  Hypokalemia: Grade 2 | 7
  Hypokalemia: Grade 4 | 1
  Hypomagnesemia: Grade 1 | 2
  Hyponatremia: Grade 1 | 15
  Hyponatremia: Grade 3 | 1
  Hypophosphatemia: Grade 1 | 4
  Hypophosphatemia: Grade 2 | 8
  Lipase increased: Grade 1 | 8
  Lipase increased: Grade 3 | 3
  Serum amylase increased: Grade 1 | 5
  Serum amylase increased: Grade 2 | 1
  Serum amylase increased: Grade 3 | 1

4. Secondary Outcome: Time to Disease Progression (TTP)
Description: TTP as assessed by investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, was define as time (in months) from date of first dose of study drug to date of first documentation of progressive disease (PD) or data censoring date, whichever occurred first. PD was defined as greater than or equal to (>=) 20 percent (%) increase in sum of diameters of target lesions, taking as a reference smallest sum on study treatment (this included baseline sum if that was smallest on study treatment), with a minimum absolute increase of at least 5 millimeter (mm), or appearance of >=1 new lesions. TTP was analyzed by Kaplan-Meier method. TTP data was censored on the date the last adequate tumor assessment for participants without PD, for participants who start new anti-cancer treatment prior to PD, for participants who died without PD, or for participants with PD after >=2 missing tumor assessments.
Time Frame: From first dose of study drug until first documentation of progressive disease or data censoring date, whichever occurred first (maximum up to 20 months)
Population: Full analysis set included all participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 22
Months | 5.52 [1.91 to 7.39]

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS as assessed by investigator per RECIST v1.1, was defined as time (in months) from date of first dose of study drug to date of first documentation of PD or death due to any cause or data censoring date, whichever occurred first. PD: >= 20% increase in sum of diameters of target lesions, taking as a reference smallest sum on study treatment (this included baseline sum if that was smallest on study treatment). The sum must also demonstrate absolute increase of >=5 mm, or appearance of >=1 new lesions. PFS was analyzed by Kaplan-Meier method. PFS data was censored on the date the last adequate tumor assessment for participants without an event (PD or death), for participants who started new anti-cancer treatment prior to PFS event, for participants with a PFS event after >=2 missing tumor assessments.
Time Frame: From first dose of study drug until first documentation of PD or death due to any cause or data censoring date, whichever occurred first (maximum up to 20 months)
Population: Full analysis set included all participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 22
Months | 5.52 [1.91 to 7.39]

6. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: OR as assessed by investigator per RECIST v.1.1, was defined as participants with confirmed best overall response of complete response (CR) or partial response (PR), were recorded from first dose of study drug until disease progression or death due to any cause. CR was defined as disappearance of all target and non-target lesions, and sustained for at least 4 weeks. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 mm. PR was defined as >=30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose of study drug until disease progression or death due to any cause (maximum up to 20 months)
Population: Full analysis set included all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 22
Percentage of participants | 13.6 [2.9 to 34.9]

7. Secondary Outcome: Percentage of Participants With Disease Control (DC)
Description: Disease control as assessed by investigator according to RECIST v1.1, was defined as participants with CR, PR, stable disease (SD), or non-CR/non-PD. CR: disappearance of all target and non-target lesions and sustained for 4 weeks. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: >= 30% decrease in sum of diameters of target lesions taking as reference baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. The sum must also demonstrate an absolute increase of at least 5 mm or appearance of >=1 new lesions. Non-CR/non-PD: Persistence of any non-target lesions and/or tumor marker level above the normal limit at >=8 weeks after date of first dose of study treatment.
Time Frame: From first dose of study drug until first documentation of CR or PR or SD or till non-CR/non-PD (maximum up to 20 months)
Population: Full analysis set included all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 22
Percentage of participants | 68.2 [45.1 to 86.1]

8. Secondary Outcome: Time to Tumor Response (TTR)
Description: TTR as assessed by investigator according to RECIST v1.1 was defined as the time (in months) from the date of first dose of study drug to the first documentation of objective response (CR or PR) that was subsequently confirmed. CR was defined as disappearance of all target and non-target lesions, and sustained for at least 4 weeks. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: >= 30% decrease in sum of diameter of target lesions taking as reference baseline sum diameters.
Time Frame: From first dose of study drug until first documentation of CR or PR (maximum up to 20 months)
Population: Full analysis set included all participants who received at least one dose of study drug.
Measure: Median (Full Range); unit: Months
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 22
Months | 1.91 [1.9 to 3.7]

9. Secondary Outcome: Duration of Response (DR)
Description: DR as assessed by investigator according to RECIST v1.1, was defined as the time from date of first documentation of objective response (CR or PR) to date of PD or death due to any cause, or data censoring date, whichever occurred first. CR: disappearance of all target and non-target lesions, and sustained for at least 4 weeks. Any pathological lymph nodes (target or non-target) reduced in short axis to <10 mm. PR: >= 30% decrease in sum of diameter of target lesions taking as reference baseline sum diameters. PD: at least a 20% increase in sum of diameters of target lesions, taking as reference the smallest sum on study treatment, with absolute increase of at least 5 mm or appearance of >=1 new lesions. DR data was censored on the date of last adequate tumor assessment for participants without an event (CR, PR, PD or death), for participants who start new anti-cancer treatment prior to DR assessment, for participants with DR assessment after >=2 missing tumor assessments.
Time Frame: From first documentation of CR or PR until first documentation of tumor progression or death due to any cause or data censoring date, whichever occurred first (maximum up to 20 months)
Population: Full analysis set included all participants who received at least one dose of study drug. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 3
Months | 7.29 [3.71 to 12.94]

10. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time (in months) from the date of first dose of study drug to the date of death due to any cause or data censoring date, whichever occurred first. Participants last known to be alive were censored at the date of last contact. OS was analyzed by Kaplan-Meier method.
Time Frame: From first dose of study drug to date of death from any cause or data censoring date, whichever occurred first (maximum up to 21 months)
Population: Full analysis set included all participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 22
Months | 14.05 [7.95 to NA] — Upper limit of 95% confidence interval (CI) could not be estimated due to low number of participants with event.

11. Secondary Outcome: Maximum Observed Serum Concentration of Avelumab
Time Frame: Pre-dose, at the end of avelumab infusion on Day 1 of Cycle 2, 3, 4 (Duration of each cycle=14 days)
Population: Pharmacokinetic (PK) analysis set included all participants who had received at least one dose of study drug and who had at least one of the PK parameters of interest for avelumab. Here, "number analyzed" signifies participants evaluable for specific time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 22
Microgram per milliliter
  Cycle 2 Day 1: number analyzed (Participants) | 21
  Cycle 2 Day 1 | 231.06 (24)
  Cycle 3 Day 1 | 228.48 (25)
  Cycle 4 Day 1: number analyzed (Participants) | 16
  Cycle 4 Day 1 | 245.66 (26)

12. Secondary Outcome: Maximum Observed Plasma Concentration of Axitinib
Time Frame: Pre-dose, 2 hours post dose Axitinib administration on Day 1 of Cycle 2, 3 (Duration of each cycle=14 days)
Population: PK analysis set included all participants who had received at least one dose of study drug and who had at least one of the PK parameters of interest for axitinib. Here, "number analyzed" signifies participants evaluable for specific time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 18
Nanograms per milliliter
  Cycle 2 Day 1 | 89.70 (23.015)
  Cycle 3 Day 1: number analyzed (Participants) | 16
  Cycle 3 Day 1 | 109.00 (17.275)

13. Secondary Outcome: Pre-dose Serum Concentration of Avelumab
Time Frame: Pre-dose on Day 1 of Cycle 2, 3, 4, 6, 8, 12, 16, 20, 24, 28 (Duration of each cycle=14 days)
Population: PK analysis set included all participants who had received at least one dose of study drug and who had at least one of the PK parameters of interest for avelumab. Here, "number analyzed" signifies participants evaluable at specific time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 22
Microgram per milliliter
  Cycle 2 Day 1 | 33.80 (17.722)
  Cycle 3 Day 1: number analyzed (Participants) | 21
  Cycle 3 Day 1 | 19.419 (64)
  Cycle 4 Day 1: number analyzed (Participants) | 17
  Cycle 4 Day 1 | 19.220 (118)
  Cycle 6 Day 1: number analyzed (Participants) | 16
  Cycle 6 Day 1 | 23.922 (68)
  Cycle 8 Day 1: number analyzed (Participants) | 13
  Cycle 8 Day 1 | 24.814 (39)
  Cycle 12 Day 1: number analyzed (Participants) | 10
  Cycle 12 Day 1 | 29.832 (37)
  Cycle 16 Day 1: number analyzed (Participants) | 9
  Cycle 16 Day 1 | 35.388 (35)
  Cycle 20 Day 1: number analyzed (Participants) | 7
  Cycle 20 Day 1 | 31.211 (36)
  Cycle 24 Day 1: number analyzed (Participants) | 5
  Cycle 24 Day 1 | 30.070 (43)
  Cycle 28 Day 1: number analyzed (Participants) | 2
  Cycle 28 Day 1 | 35.578 (19)

14. Secondary Outcome: Pre-dose Plasma Concentration of Axitinib
Time Frame: Pre-dose on Day 1 of Cycle 2 and 3 (Duration of each cycle=14 days)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 18
Nanograms per milliliter
  Cycle 2 Day 1 | 11.6439 (123)
  Cycle 3 Day 1: number analyzed (Participants) | 16
  Cycle 3 Day 1 | 9.2226 (164)

15. Secondary Outcome: Number of Participants With Their Target Programmed Death-Ligand 1 (PD-L1) Status
Description: PD-L1 status was defined as positive when PD-L1 staining of any intensity was observed in tumor-associated immune cells covering >= 1% of the tumor area. PD-L1 status was defined as negative when PD-L1 staining of any intensity was observed in tumor-associated immune cells covering < 1% of the tumor area.
Time Frame: Baseline (Day 1)
Population: PD-L1 biomarker analysis set included participants who had received at least one dose of study drug and who had at least one screening biomarker assessment for PD-L1.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 20
Participants
  PD-L1: Positive | 17
  PD-L1: Negative | 3

16. Secondary Outcome: Mean Percentage of CD8+ Cells in Per Unit Area of Invasive Margin, Center of Tumor Cells and Total Area of Tumor Cells
Description: CD8+ cells are the type of T-lymphocytes. Invasive margin is defined as the region on each side of the border between tumor cells. Expression of CD8+ cells in invasive margin, center of tumor cells, total area of tumor cells has been reported as mean percentage of CD8+cells per unit area. Area was measured in millimeter square (mm^2).
Time Frame: From first dose of study drug up to end of treatment (maximum up to 20 months)
Population: CD8+ biomarker analysis set included participants who had received at least one dose of study drug and who had at least one screening biomarker assessment for CD8+ cells. Here, "number analyzed" signifies participants evaluable for specific rows.
Measure: Mean (Standard Deviation); unit: Percentage of CD8+cells per mm^2
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 20
Percentage of CD8+cells per mm^2
  CD8+ Cells in Invasive Margin: number analyzed (Participants) | 7
  CD8+ Cells in Invasive Margin | 2.12 (1.760)
  CD8+ Cells in Center of Tumor Cells: number analyzed (Participants) | 19
  CD8+ Cells in Center of Tumor Cells | 0.91 (1.328)
  CD8+ Cells in Total Area of Tumor Cells: number analyzed (Participants) | 19
  CD8+ Cells in Total Area of Tumor Cells | 1.02 (1.353)

17. Secondary Outcome: Summary of Cluster of Differentiation 8 (CD8+) Cells Expression: Total Area Covered by CD8+ Cells in Center of Tumor Cells
Description: CD8+ cells are the type of T-lymphocytes.
Time Frame: From first dose of study drug up to end of treatment (up to 20 months)
Population: CD8+ biomarker analysis set included participants who had received at least one dose of study drug and who had at least one screening biomarker assessment for CD8+ cells. Here, "Overall Number of Participants Analyzed" signifies the number of participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 19
mm^2 | 53.88 (48.832)

18. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADAs) and Positive Neutralizing Antibodies (nAbs)
Description: ADA positive was defined as presence of at least one positive ADA sample. nAb positive was defined as presence of at least one positive nAb sample.
Time Frame: From first dose of study drug until 30 days after the last dose of study drug (maximum up to 21 months)
Population: The immunogenicity analysis set included participants who have received at least one dose of study drug and who had at least one ADA or nAb sample collected for avelumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 22
Participants
  ADA positive | 3
  nAb positive | 3

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after last dose of study drug or initiation of new anti-cancer drug therapy, whichever occurred first (maximum up to 21 months)
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Avelumab + Axitinib
All-Cause Mortality (participants affected / at risk) | 12/22
Serious Adverse Events (participants affected / at risk) | 8/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab + Axitinib (N=22)
Acute myocardial infarction (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Malaise (General disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Headache (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab + Axitinib (N=22)
Adrenal insufficiency (Endocrine disorders) | 2
Hyperthyroidism (Endocrine disorders) | 3
Hypothyroidism (Endocrine disorders) | 7
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 3
Anal erosion (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 6
Glossitis (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 3
Malaise (General disorders) | 7
Oedema (General disorders) | 2
Oedema peripheral (General disorders) | 4
Pyrexia (General disorders) | 6
Nasopharyngitis (Infections and infestations) | 4
Paronychia (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 3
Contusion (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Platelet count decreased (Investigations) | 2
Transaminases increased (Investigations) | 2
Weight decreased (Investigations) | 9
Decreased appetite (Metabolism and nutrition disorders) | 12
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Dysgeusia (Nervous system disorders) | 6
Headache (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 3
Haematuria (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 11
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 6
Hypertension (Vascular disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-05-18): https://cdn.clinicaltrials.gov/large-docs/33/NCT03289533/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT03289533/SAP_001.pdf